CLINICAL TRIAL: NCT00215709
Title: A Pilot Study of Docetaxel on a Bi-Weekly Schedule in the Treatment of Elderly Men With Hormone-Refractory Prostate Cancer (HRPC)
Brief Title: Bi-Weekly Administration of Docetaxel for Older Men With Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Geriatric Oncology Consortium (Other)
Collaborators: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOC GU-010
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-11

CONDITIONS: Prostate Cancer
Keywords: elderly
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: docetaxel

SUMMARY:
This pilot study is designed to determine the feasibility and safety of administering docetaxel at various dosing levels on a bi-weekly schedule in older men with hormone refractory prostate cancer.

DETAILED DESCRIPTION:
The information obtained from this trial will help determine the feasibility and safety of administering docetaxel at various dosing levels on a bi-weekly schedule in this patient population. If the data from this phase I trial are encouraging, a phase II trial will be conducted to further assess the efficacy of this dosing schedule.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 65 years;
* histologically confirmed adenocarcinoma of the prostate;
* metastatic disease;
* unresponsive or refractory to hormonal therapy, as defined by at least 1 of the following criteria: progression of bidimensionally measurable disease; progression of evaluable but not measurable disease (bone scan); at least 2 consecutive rises in PSA at least 1 week apart;
* patients must have serum testosterone levels < 50 ng/mL at time of study entry. For patients who are medically castrated, lutenizing hormone releasing hormone analog must continue to maintain testicular suppression;
* prior nonsteroidal antiandrogens (flutamide, ketoconazole, bicalutamide, or nilutamide) allowed if disease progression occurred. No evidence of response after antiandrogen withdrawal within 4 weeks for patients treated with flutamide, ketoconazole, nilutamide and 6 weeks for patients treated with bicalutamide;
* chemotherapy naïve;
* full recovery from the effects of any prior surgery or radiation therapy. At least 4 weeks since any radiation therapy;
* ECOG performance status 0-2;
* adequate kidney, liver, and bone marrow functions;
* signed study-specific informed consent form.

Exclusion Criteria:

* Concurrent chemotherapy or immunotherapy;
* Patients who have received an investigational drug within 4 weeks of registration;
* Prior or concurrent malignancies (other than surgically treated carcinoma in situ of the cervix and squamous or basal cell carcinoma of the skin) within the preceding five years;
* Serious medical or psychiatric illness which would prevent informed consent;
* Life expectancy < 3 months;
* Active uncontrolled bacterial, viral, or fungal infection until these conditions are corrected or controlled;
* Known hypersensitivity to study drug or to other drugs formulated with polysorbate 80.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-07; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of docetaxel on a bi-weekly schedule in the treatment of elderly men with hormonal refractory prostate cancer (HRPC).

SECONDARY OUTCOMES:
To determine the dose limiting toxicity effects and other toxic effects of this regimen
To determine the activity of this regimen in terms of: Overall response rates; Pain scores and analgesic use; PSA response rates;
To evaluate the feasibility of using a self-report geriatric assessment tool in this population

CONTACTS AND LOCATIONS:
Overall Officials: William Ershler, MD, Principal Investigator — Geriatric Oncology Consortium
Locations (1):
- Baltimore, Maryland, United States

REFERENCES:
- See also: Geriatric Oncology Consoritum website — http://www.thegoc.org